CLINICAL TRIAL: NCT01597180
Title: Pharmacokinetics, Pharmacodynamics and Genital Tract Viral Shedding in HIV+ Women Using Combined Oral Contraceptives and Raltegravir
Brief Title: Pharmacokinetics, Pharmacodynamics and Cervicovaginal Lavage of Combined Oral Contraceptives and Raltegravir
Status: Withdrawn | Type: Observational
Why Stopped: Could not find subjects who met all the enrollment criteria so the study was stopped.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gretchen Stuart, MD, Associate Professor, Department of Obstetrics and Gynecology, University of North Carolina, Chapel Hill
Other Study IDs: 12-0832
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: HIV
Keywords: contraception; HIV; pharmacokinetics; pharmacodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to learn about potential interactions between raltegravir and a birth control pill in HIV+ women. The investigators plan to enroll HIV+ women who are on steady state raltegravir containing highly active antiretroviral therapy (HAART), ages 20-40, inclusive, who report regular monthly menses.

The investigators will investigate drug interactions of raltegravir, ethinyl estradiol (EE) and levonorgestrel (LNG). All women will be receiving raltegravir as part of their regular medical care. Women will be enrolled in the study for approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20-40 years of age with regular monthly menses
* If over age 35 then must not use tobacco
* Negative pregnancy test
* No known allergy to raltegravir
* No known history of phenylketonuria
* Undetectable HIV viral load
* No active liver disease as determined by medical history and normal AST and ALT
* No history of hepatic adenomas, carcinomas or benign liver tumors
* Ho history of thrombophlebitis of thromboembolic disease
* No history of deep vein thrombosis
* No history of cerebral vascular or coronary artery disease
* No known or suspected carcinoma of the breast
* No undiagnosed abnormal genital bleeding
* Not taking concomitant CYP 450 inducing medications such as anti-seizure medications
* No use of oral contraceptives, depot-medroxyprogesterone acetate, contraceptive ring or patch within two months of screening
* No cholestatic jaundice of pregnancy or jaundice with prior contraceptive pill use
* Has used raltegravir prior to screening
* Has no history of malignancy of the genital tract (e.g. cervical cancer, ovarian cancer, endometrial cancer)
* Must not have had an abnormal pap test defined without resolution in the last 18 months.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women recruited from an infectious diseases clinic in Chapel Hill, NC.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in cervicovaginal fluide milieu

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen S Stuart, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Infectious Disease Clinic, Chapel Hill, North Carolina, United States